CLINICAL TRIAL: NCT02729025
Title: A RaNdomized Double-blInd Placebo ConTrolled Study Characterizing THe Effects of PCSK9 Inhibition On Arterial Wall Inflammation in Patients With Elevated Lp(a) (ANITSCHKOW)
Brief Title: Effects of Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9) Inhibition on Arterial Wall Inflammation in Patients With Elevated Lipoprotein(a) (Lp(a))
Acronym: ANITSCHKOW
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20130293; 2015-003731-35 (EudraCT Number)
Record Dates: First submitted 2016-03-08; First posted 2016-04-06 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Subjects With Hyperlipidemia, Dyslipidemia
Keywords: Hyperlipidemia; Dyslipidemia; Proprotein convertase subtilisin/kexin type 9 (PCSK9) Inhibition; Arterial Wall Inflamation; Elevated lipoprotein a
MeSH Terms: conditions — Dyslipidemias; Hyperlipidemias; Hypercholesterolemia, Autosomal Dominant, 3; Inhibition, Psychological | interventions — evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo to evolocumab by subcutaneous injection once a month (QM) for 12 weeks.
  Interventions: Drug: Placebo
- Evolocumab 420 mg QM (Experimental): Participants received 420 mg evolocumab by subcutaneous injection once a month (QM) for 12 weeks.
  Interventions: Drug: Evolocumab

INTERVENTIONS:
Drug: Evolocumab — Administered subcutaneously once a month using an autoinjector/pen.
  Other Names: Repatha; AMG 145
  Arms: Evolocumab 420 mg QM
Drug: Placebo — Administered subcutaneously once a month using an autoinjector/pen.
  Arms: Placebo

SUMMARY:
A study to assess the effects of proprotein convertase subtilisin/ kexin type 9 (PCSK9) inhibition on the arterial wall inflammation in patients with elevated lipoprotein(a).

ELIGIBILITY:
Inclusion Criteria:

* Fasting lipoprotein(a) (Lp(a)) 50 mg/dL or more at screening 1
* Fasting Low-density lipoprotein-cholesterol (LDL-C) 100 mg/dL or more at screening 1
* Lipid lowering therapy including statin dose unchanged for at least 8 weeks prior to screening
* Target-to-background ratio (TBR) maximum higher than 1.6 (either right, left carotid or thoracic aorta) on fluorodeoxyglucose-positron emission tomography/computed tomography (FDG-PET/CT).

Exclusion Criteria:

* Currently receiving, or less than 4 weeks since receiving, treatment in another investigational device or drug study(ies), or participating in other investigational procedures
* Known diagnosis of diabetes mellitus or screening fasting serum glucose ≥ 126 mg/dL or hemoglobin A1C (HbA1C) ≥ 6.5%
* Subject with a history of homozygous familial hypercholesterolemia
* History of a Cardiovascular event
* Subject currently undergoing lipid apheresis
* Known contraindications or limitations to FDG-PET/ CT (scanner weight limit, devices that can cause image artifacts, or carotid/aortic stents/grafts
* Subject has had exposure to investigational drugs targeting Lp(a) within the last 12 months, prior to Screening
* Other Exclusion Criteria May Apply.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2018-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (15):
- United States (5):
  - Research Site, Miami, Florida
  - Research Site, Las Vegas, Nevada
  - Research Site, Mooresville, North Carolina
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Hurst, Texas
- Canada (4):
  - Research Site, Newmarket, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Québec, Quebec
- Netherlands (6):
  - Research Site, Amsterdam
  - Research Site, Apeldoorn
  - Research Site, Nijmegen
  - Research Site, Rotterdam
  - Research Site, Venlo
  - Research Site, Waalwijk

REFERENCES:
- [Background] Stiekema LCA, Stroes ESG, Verweij SL, Kassahun H, Chen L, Wasserman SM, Sabatine MS, Mani V, Fayad ZA. Persistent arterial wall inflammation in patients with elevated lipoprotein(a) despite strong low-density lipoprotein cholesterol reduction by proprotein convertase subtilisin/kexin type 9 antibody treatment. Eur Heart J. 2019 Sep 1;40(33):2775-2781. doi: 10.1093/eurheartj/ehy862. PMID 30561610
- [Derived] Schmidt AF, Carter JL, Pearce LS, Wilkins JT, Overington JP, Hingorani AD, Casas JP. PCSK9 monoclonal antibodies for the primary and secondary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2020 Oct 20;10(10):CD011748. doi: 10.1002/14651858.CD011748.pub3. PMID 33078867
- [Derived] Zhang X, Stiekema LCA, Stroes ESG, Groen AK. Metabolic effects of PCSK9 inhibition with Evolocumab in subjects with elevated Lp(a). Lipids Health Dis. 2020 May 11;19(1):91. doi: 10.1186/s12944-020-01280-0. PMID 32393252
- [Derived] Stiekema LCA, Prange KHM, Hoogeveen RM, Verweij SL, Kroon J, Schnitzler JG, Dzobo KE, Cupido AJ, Tsimikas S, Stroes ESG, de Winther MPJ, Bahjat M. Potent lipoprotein(a) lowering following apolipoprotein(a) antisense treatment reduces the pro-inflammatory activation of circulating monocytes in patients with elevated lipoprotein(a). Eur Heart J. 2020 Jun 21;41(24):2262-2271. doi: 10.1093/eurheartj/ehaa171. PMID 32268367
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 14 centers in Canada, the Netherlands, and the United States. Participants were enrolled from 14 April 2016 to 07 December 2017.
Pre-assignment Details: Eligible participants were randomized in a 1:1 ratio to receive either evolocumab or placebo. Randomization was stratified by baseline background statin therapy (on statin versus not on statin) and by screening lipoprotein(a) (Lp[a]) (< 175 mg/dL or ≥ 175 mg/dL).
Period: Overall Study
Arm/Group | Placebo | Evolocumab 420 mg QM
Started | 64 | 65
Completed | 64 | 64
Not Completed | 0 | 1
Not completed — Sponsor Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Evolocumab 420 mg QM | Total
Number analyzed (Participants) | 64 | 65 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (7.6) | 60.0 (6.8) | 60.3 (7.2)
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 41 | 48 | 89
  ≥ 65 years | 23 | 17 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 39 | 69
  Male | 34 | 26 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 64 | 64 | 128
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Black or African American | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 58 | 58 | 116
  Other | 0 | 1 | 1
Location of the Index Vessel Used for Calculation of Maximum Target-to-background Ratio [Count of Participants; unit: Participants] — The index vessel used to calculate the mean of the maximum target-to-background ratio in the most diseased segment at baseline. Using quantitative fluorodeoxyglucose-positron emission tomography/computed tomography (FDG-PET/CT) image analysis, the artery (right carotid, left carotid, or thoracic aorta) with the highest FDG uptake (highest mean of the maximum target-to-background ratio at baseline) was identified as the index vessel.
  Participants
    Ascending thoracic aorta | 54 | 49 | 103
    Left common carotid | 1 | 3 | 4
    Right common carotid | 8 | 11 | 19
    Missing | 1 | 2 | 3
Maximum Target-to-background Ratio (TBR) in the Most Diseased Section of the Index Vessel [Mean (Standard Deviation); unit: ratio] — Arterial inflammation was assessed using 18F-fluoro-deoxyglucose positron-emission tomography/computed tomography (18F-FDG PET/CT).
  Maximum standardized uptake was calculated as a time- and dose- corrected tissue radioactivity divided by body weight in the index vessel and TBR was calculated from the ratio of the standardized uptake value of the artery compared to mean background venous activity. Maximum TBR for the most diseased segment (MDS) was calculated from a group of 3 contiguous slices (approximately 1.5 cm), centered on the slice with the highest maximum TBR in the index vessel. Population: Participants with available data
  ratio
    number analyzed (Participants) | 63 | 63 | 126
    (all) | 2.28765 (0.41284) | 2.29667 (0.46063) | 2.29216 (0.43566)
Stratification Factor: Baseline Statin Therapy [Count of Participants; unit: Participants]
  Yes | 33 | 34 | 67
  No | 31 | 31 | 62
Stratification Factor: Screening Lipoprotein(a) (Lp[a]) Level [Count of Participants; unit: Participants]
  < 175 mg/dL | 60 | 61 | 121
  ≥ 175 mg/dL | 4 | 4 | 8
Lipoprotein(a) Concentration [Median (Inter-Quartile Range); unit: nmol/L] | 198.0 [151.3 to 300.0] | 203.0 [162.5 to 301.5] | 200.0 [155.5 to 301.5]
Low-density Lipoprotein Cholesterol (LDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] | 141.7 (35.7) | 146.2 (43.5) | 144.0 (39.7)
Apolipoprotein B Concentration [Mean (Standard Deviation); unit: mg/dL] | 108.0 (22.9) | 109.9 (23.7) | 108.9 (23.2)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Maximum Target-to-background Ratio in the Most Diseased Segment of the Index Vessel at Week 16
Description: Arterial inflammation was assessed using 18F-fluoro-deoxyglucose positron-emission tomography/computed tomography (18F-FDG PET/CT). Arterial 18F-FDG uptake is correlated with arterial macrophage content and predicts cardiovascular events. Images were analyzed by an experienced radiologist blinded to all patient characteristics.
  The maximum standardized uptake value was calculated as a time- and dose- corrected tissue radioactivity divided by body weight in the index and the target-to-background ratio (TBR) was calculated from the ratio of the standardized uptake value of the artery compared to mean background venous activity. The average maximum TBR for the most diseased segment (MDS) was calculated from a group of 3 contiguous slices (approximately 1.5 cm), centered on the slice with the highest maximum TBR in the index vessel. The index vessel was defined as the vessel (either the right or left carotid or aorta) with the highest mean TBR at baseline.
Time Frame: Baseline and week 16
Population: Participants who received at least 1 dose of study drug with available data
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab 420 mg QM
Number analyzed (Participants) | 63 | 63
percent change | -5.31 (1.67) | -8.31 (1.67)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab 420 mg QM; A multivariate regression was modelled on the primary endpoint as well as three other response variables (percent change in Lp[a] at Weeks 8 and 16, baseline MDS TBR, and baseline Lp[a]). The primary endpoint was regressed on the treatment group and statin stratification factor; baseline MDS TBR and Lp(a) were regressed on the statin stratification factor, and percent changes in Lp(a) were regressed on the treatment group, statin stratification factor, visit, and treatment group by visit; Test type: Superiority; p = 0.18, Multivariate regression model; LS Mean Treatment Difference = -3.00, 95% CI 2-sided [-7.40 to 1.39], Standard Error of Mean 2.24 — Treatment difference used placebo as the reference

2. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) Concentration at Week 16
Time Frame: Baseline and week 16
Population: Participants who received at least 1 dose of study drug with available data
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab 420 mg QM
Number analyzed (Participants) | 61 | 63
percent change | 1.06 (1.94) | -12.83 (1.92)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab 420 mg QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model; The model included treatment group, statin stratification, scheduled visit, and the interaction of treatment with scheduled visit; LS Mean Treatment Difference = -13.89, 95% CI 2-sided [-19.29 to -8.49], Standard Error of Mean 2.73 — Treatment difference used placebo as the reference

3. Secondary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C) Concentration at Week 16
Time Frame: Baseline and week 16
Population: Participants who received at least 1 dose of study drug with available data
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab 420 mg QM
Number analyzed (Participants) | 59 | 62
percent change | 1.64 (1.86) | -59.02 (1.82)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab 420 mg QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model; [statistical method as in outcome 2, analysis 1]; LS Mean Treatment Difference = -60.66, 95% CI 2-sided [-65.81 to -55.51], Standard Error of Mean 2.60 — Treatment difference used placebo as the reference

4. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B Concentration at Week 16
Time Frame: Baseline and week 16
Population: Participants who received at least 1 dose of study drug with available data
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab 420 mg QM
Number analyzed (Participants) | 61 | 63
percent change | 3.29 (1.53) | -48.30 (1.51)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab 420 mg QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model; [statistical method as in outcome 2, analysis 1]; LS Mean Treatment Difference = -51.29, 95% CI 2-sided [-55.85 to -47.33], Standard Error of Mean 2.15 — Treatment difference used placebo as the reference

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 30 days after the last dose or until the end of study date, whichever was earlier; the maximum duration of treatment was 3.9 months.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Placebo QM: Participants received placebo to evolocumab by subcutaneous injection once a month (QM) for 12 weeks.
Arm/Group | Placebo QM | Evolocumab 420 mg QM
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/64 | 2/65
Other Adverse Events (participants affected / at risk) | 47/64 | 49/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo QM (N=64) | Evolocumab 420 mg QM (N=65)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo QM (N=64) | Evolocumab 420 mg QM (N=65)
Palpitations (Cardiac disorders) | 0 | 1
Dermoid cyst (Congenital, familial and genetic disorders) | 1 | 0
Muscular dystrophy (Congenital, familial and genetic disorders) | 1 | 0
Excessive cerumen production (Ear and labyrinth disorders) | 1 | 0
Keratitis (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 5 | 1
Oesophageal pain (Gastrointestinal disorders) | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 3 | 0
Chills (General disorders) | 0 | 1
Drug intolerance (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 2
Influenza like illness (General disorders) | 4 | 4
Injection site hypersensitivity (General disorders) | 1 | 0
Injection site pain (General disorders) | 1 | 1
Injection site rash (General disorders) | 1 | 0
Nodule (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 1
Bronchitis (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1
H1N1 influenza (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Heterophyiasis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 3 | 7
Nail infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 13 | 6
Otitis externa (Infections and infestations) | 0 | 1
Root canal infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 3 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Bone contusion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 0
Weight decreased (Investigations) | 1 | 1
Weight increased (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 3
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 3
Headache (Nervous system disorders) | 7 | 4
Hypoaesthesia (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 1
Memory impairment (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 2 | 1
Retinal migraine (Nervous system disorders) | 1 | 0
Speech disorder (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 4
Irritability (Psychiatric disorders) | 0 | 1
Menopausal symptoms (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1
Bunion operation (Surgical and medical procedures) | 1 | 0
Flushing (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 3
Peripheral coldness (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2017-02-08): https://cdn.clinicaltrials.gov/large-docs/25/NCT02729025/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/25/NCT02729025/SAP_001.pdf